CLINICAL TRIAL: NCT03933046
Title: The Association Between Sleep Duration and Sleep Disorders and Proteinuria in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0134-19-TLV
Record Dates: First submitted 2019-04-14; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: OSA; Proteinuria; Periodic Limb Movement Sleep Disorder
Keywords: osa; proteinuria; periodic limb movement disorder; children
MeSH Terms: conditions — Proteinuria; Sleep Apnea, Obstructive; Nocturnal Myoclonus Syndrome | interventions — Urinalysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children referred to PSG due to suspected SDB (Experimental)
  Interventions: Diagnostic Test: PSG

INTERVENTIONS:
Diagnostic Test: PSG — polysomnography and urine analaysis for protein levels
  Other Names: urine analysis

SUMMARY:
The presence of protein in urine is a common laboratory finding in children. Although proteinuria is usually benign, it can be a marker of a serious underlying renal disease or systemic disorder. Microalbuminuria can be one of the first subclinical manifestations of endothelial dysfunction and is associated with low grade systemic inflammation. Multiple studies from the adult population suggest that microalbuminuria above the upper quartile is linked with increased risk of coronary heart disease and death even after adjustment for the presence of diabetes mellitus, obesity and hypertension.

Obstructive sleep apnea (OSA) has been recognized as an independent risk factor for cardiovascular morbidity related to sympathetic nervous system overflow, metabolic dysregulation, inflammation and endothelial dysfunction secondary to repetitive hypoxia -reoxygenation events.

Therefore, there is a need for further studies to investigate the association between OSA and microalbuminuria in children. Furthermore, no studies have thus far investigated the association between other sleep disorders such as periodic limb movement (PLMD) and microalbuminuria in children.

Our hypothesis is that children with sleep disorders or short sleep duration have increased risk of proteinuria/microalbuminuria and that treatment and resolution of the sleep problem will be followed by improvement in proteinuria levels.

DETAILED DESCRIPTION:
200 children aged 2-18 years that will be referred to the Sleep Disorders Center for overnight polysomnography due to suspected sleep disordered breathing or PLMD will be recruited to the study during their first visit in the sleep clinic. During that study, an informed consent will be completed by the parents. Data on weekdays and weekends sleep duration as well as personal and family history of kidney disease will be collected.

Exclusion criteria:1. Known renal disease; 2. diabetes mellitus; 3. current use of ACE inhibitors or angiotensin receptor blockers; 4. neuromuscular disorders or craniofacial abnormalities; 5. syndromic conditions.

All participants will undergo physical examination. Weight and height will be measured, and body mass index (BMI) z-score will be calculated.

Blood pressure will be measured on the first visit in the sleep clinic by a trained physician as specified in recent guidelines. 19

Overnight polysomnography will be carried out in the Sleep Disorders Laboratory and the following signals will be recorded: electroencephalogram (EEG; C3/M2, C2/M1, O1/M2, O2/M1); right and left oculogram; submental and tibial electromyogram; body position; electrocardiogram; thoracic and abdominal wall motion; oronasal airflow (three-pronged thermistor and nasal pressure transducer); and oxygen saturation of hemoglobin (SpO2). Arousals, sleep stages and respiratory events will be scored, and polysomnography indices will be defined according to the recent American Academy of Sleep Medicine recommendations . 20

First void urine samples will be collected in a sterile cup the morning following the polysomnography (6:00-7:00 am). For each sample urinalysis, protein/creatinine and albumin/creatinine will be measured. Urinary albumin and protein excretion will be the primary outcome measure. Proteinuria will be defined as protein/creatinine greater than 0.2 and albuminuria will be defined as albumin/creatinine above age-adjusted limits Children who will be diagnosed with moderate-severe OSA will be referred to an ENT surgeon for adenotonsillectomy, the first line of treatment in pediatric OSA. Six to 10 weeks following surgery, these children will be requested to undergo additional PSG evaluation. First void urine samples will be collected the following morning.

In addition- 100 children referred to the pediatric nephrology clinic due to asymptomatic albuminuria/proteinuria will be recruited. Parents will be required to complete a designated sleep questionnaire that includes items on sleep duration, SDB and RLS symptoms. Exclusion criteria, as described above for the entire cohort, will also apply to this subpopulation.

Informed consent will be completed by the parents.

ELIGIBILITY:
Inclusion Criteria:

1. age: 2-17 years
2. Referred to overnight PSG due to suspected OSA or PLMD
3. referred for evaluation in the nephrology clinic due to proteinuria

Exclusion Criteria:

1. Known renal disease;
2. diabetes mellitus;
3. current use of ACE inhibitors or angiotensin receptor blockers;
4. neuromuscular disorders
5. craniofacial abnormalities
6. syndromic conditions.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
morning urine protein/creatinine >0.2 | 1 year
reported sleep duration (hours) | 1 year
morning urine protein/creatinine >0.2 post treatment of OSA | 1 year